CLINICAL TRIAL: NCT06737575
Title: Validation of Chest Trauma Scoring Systems in Predicting Blunt Chest Injury Outcomes in Iraq: A Prospective Study
Brief Title: Chest Trauma Scoring Systems as Predictors of Morbidity and Mortality in Iraq
Acronym: CTS
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241212A; 013 (Other: Nahrain Medical Research Collective (NMRC))
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Chest Injury Trauma Blunt
Keywords: CTS; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This prospective observational study aims to evaluate the effectiveness of chest trauma scoring systems in predicting morbidity and mortality in patients with blunt chest trauma in Iraq. The primary questions it seeks to address are:

How accurately do chest trauma scoring systems predict mortality and critical outcomes such as ICU admission or the need for advanced interventions? How well do these scoring systems stratify patients based on injury severity in a resource-limited setting? Are there any demographic or clinical factors that impact the predictive performance of these scoring systems?

Participants will:

Be assessed using chest trauma scoring systems upon arrival at the emergency department to determine risk levels.

Have demographic and clinical data, including age, gender, injury mechanism, comorbidities, and length of hospital stay, collected to explore potential associations with outcomes.

DETAILED DESCRIPTION:
Chest trauma is a major cause of morbidity and mortality, often resulting from motor vehicle accidents, falls, or physical assaults. It can lead to serious complications such as pulmonary contusions, rib fractures, and damage to thoracic organs. The Chest Trauma Score (CTS) helps assess injury severity by considering factors like age, number of rib fractures, and pulmonary contusion severity. Higher CTS values are associated with worse outcomes, such as prolonged mechanical ventilation and higher mortality rates. Early identification using this scoring system improves clinical decision-making and outcomes.

Despite the global utility of trauma scoring systems, there is limited research on their application in developing countries like Iraq, where trauma care is often constrained by limited resources and inconsistent protocols. In Iraq, blunt chest trauma is a prevalent issue due to frequent road traffic accidents and other causes. However, a lack of locally validated tools such as CTS hinders the ability of healthcare providers to assess injury severity accurately and predict outcomes.

This study aims to evaluate the effectiveness of the Chest Trauma Score in predicting morbidity and mortality among patients with blunt chest trauma in Iraq. By addressing this research gap, the findings will contribute to improving trauma care protocols, informing policy decisions, and enhancing the overall healthcare system's capacity to manage chest trauma effectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with blunt chest trauma.
* Patients presenting to the emergency department within 4 hours.
* Patients (or their legal representatives) must provide informed consent to participate in the study.
* Patients who can be assessed using the Chest Trauma Score at the time of arrival (e.g., having stable enough vitals to allow for evaluation).

Exclusion Criteria:

* Patients with penetrating chest trauma (e.g., gunshot or stab wounds), as the Chest Trauma Score is typically used for blunt trauma.
* Patients presenting with chest conditions unrelated to trauma (e.g., pneumonia, COPD exacerbation, or other non-traumatic causes of chest pain or respiratory distress).
* Patients with severe pre-existing comorbidities (e.g., end-stage heart failure, terminal cancer) where trauma is unlikely to be the primary cause of morbidity or mortality.
* Patients with missing or incomplete clinical data, including imaging or vital signs necessary to calculate the CTS accurately.
* Patients who refuse consent or do not agree to the use of their data for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients aged 18 years and older presenting to the emergency department with blunt chest trauma. Participants will be assessed using the Chest Trauma Score (CTS) to predict morbidity and mortality, and data on demographics, injury mechanisms, and clinical outcomes will be collected. The study aims to include a diverse sample from varying age groups and both genders to evaluate the score's performance across different subgroups.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | In-Hospital Phase (average of 10 days through discharge); Post-Discharge Follow-Up: Day 7, Day 30
  Mortality (death) during hospitalization.
Accuracy Assessment of the Chest Trauma Score (CTS) | the first 4 hours after ER admission
  The total score ranges from 2 to 12, with higher scores indicating worse outcomes.

SECONDARY OUTCOMES:
Number of Participants Requiring ICU Admission | Up to discharge, an average of 10 days
  The requirement for admission to the intensive care unit (ICU) is determined by the presence of severe clinical deterioration, significant complications, or the need for advanced monitoring and life-support measures.

CONTACTS AND LOCATIONS:
Overall Officials: Yaser aamer Eisa Alhaibi, Assistant professor, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Battle C, Cole E, Carter K, Baker E. Clinical prediction models for the management of blunt chest trauma in the emergency department: a systematic review. BMC Emerg Med. 2024 Oct 12;24(1):189. doi: 10.1186/s12873-024-01107-6. PMID 39395934
- [Result] Dogrul BN, Kiliccalan I, Asci ES, Peker SC. Blunt trauma related chest wall and pulmonary injuries: An overview. Chin J Traumatol. 2020 Jun;23(3):125-138. doi: 10.1016/j.cjtee.2020.04.003. Epub 2020 Apr 20. PMID 32417043